CLINICAL TRIAL: NCT04418011
Title: Neuromodulation of Social Cognitive Circuitry in People With Schizophrenia Spectrum Disorders
Acronym: ModSoCCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Northwell Health (Other); University of Maryland, Baltimore (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 133/2019
Record Dates: First submitted 2020-05-05; First posted 2020-06-05 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Active 10 Hz rTMS (Active Comparator): Active treatment will be targeted to an intensity that is 120% of the resting motor threshold. Stimulation will be delivered at 10 Hz according to conventional FDA-approved parameters (4 s on and 26 s off; 3000 pulses per session; total duration 37.5 mins) .
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Active iTBS (Active Comparator): Active iTBS will be targeted to an intensity that is 120% of the resting motor threshold. Stimulation will be delivered in triplet 50 Hz bursts, repeated at 5 Hz; 2 seconds on and 8 seconds off; 600 pulses per session; total duration of 3 min 9 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (Intermittent Theta Burst Stimulation)
- Sham rTMS (Sham Comparator): Sham stimulation will be delivered using the same stimulation parameters as either 10 Hz rTMS or iTBS.
  For both active and sham stimulation, TMS coil positioning for each individual will be optimized by combining participant fMRI data, meta-analytic functional analysis, electric field modelling, and real-time neuronavigation.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (Sham)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — The present study aims to use both repetitive transcranial magnetic stimulation (rTMS) and intermittent theta burst stimulation (iTBS), safe and effective forms of neuromodulation, to target the neural circuitry of social cognitive (SCog) impairments in people with SSDs. Treatment sessions will be administered five days per week for two weeks.
  Other Name: MagPro X100 or R30 (Medtronic A/S. Copenhagen, Denmark) equipped with a Cool-B70 A/P coil and Qooler fluid-cooling device (MagVenture, Farum, Denmark), positioned under MRI guidance using the Brainsight neuronavigation system (Rogue Resolutions, Montreal, Canada) or Localite (Localite GmbH, Bonn, Germany)
  Arms: Active 10 Hz rTMS
Device: Repetitive Transcranial Magnetic Stimulation (Intermittent Theta Burst Stimulation) — The present study aims to use both repetitive transcranial magnetic stimulation (rTMS) and intermittent theta burst stimulation (iTBS), safe and effective forms of neuromodulation, to target the neural circuitry of social cognitive (SCog) impairments in people with SSDs. Treatment sessions will be administered five days per week for two weeks.
  Other Name: MagPro X100 or R30 (Medtronic A/S. Copenhagen, Denmark) equipped with a Cool-B70 A/P coil and Qooler fluid-cooling device (MagVenture, Farum, Denmark), positioned under MRI guidance using the Brainsight neuronavigation system (Rogue Resolutions, Montreal, Canada) or Localite (Localite GmbH, Bonn, Germany)
  Arms: Active iTBS
Device: Repetitive Transcranial Magnetic Stimulation (Sham) — Other Name: MagPro X100 or R30(Medtronic A/S. Copenhagen, Denmark) equipped with a Cool-B70 A/P coil and Qooler fluid-cooling device (MagVenture, Farum, Denmark), positioned under MRI guidance using the Brainsight neuronavigation system (Rogue Resolutions, Montreal, Canada) or Localite (Localite GmbH, Bonn, Germany)
  Arms: Sham rTMS

SUMMARY:
In this study, the investigators will be examining the effects of repetitive transcranial magnetic stimulation (rTMS) and intermittent theta burst stimulation (iTBS) on social cognitive impairments in individuals with schizophrenia spectrum disorders. Participants will be chosen by chance to receive either active rTMS stimulation, active iTBS stimulation, sham rTMS, or sham iTBS. The investigators predict that active 10Hz and iTBS stimulation will improve social cognitive impairments compared to sham stimulation. We aim to identify which type of active stimulation is most effective at inducing changes social cognition brain circuitry and secondarily which type of active stimulation is best tolerated and most effective at inducing changes in social cognitive performance.

DETAILED DESCRIPTION:
This study is a randomized, double blind, sham controlled study which aims to use repetitive transcranial magnetic stimulation (rTMS), a form of neuromodulation, to target the neural circuitry of social cognitive (SCog) impairments in people with Schizophrenia Spectrum Disorders. We will randomize 60 people with SSDs to three groups: 20 to a conventional form of rTMS (i.e. 10 Hz rTMS); 20 to intermittent theta burst stimulation (iTBS); and 20 to either sham 10Hz rTMS stimulation or sham iTBS. We will determine whether these treatments can change the functional connectivity of key SCog brain circuits by targeting a brain region known as the dorsomedial prefrontal cortex (DMPFC). Since each person's anatomical and functional brain profile is slightly different, we will optimize the orientation and location of coil placement in each individual. Overall, our proposal follows a target engagement framework, including specifics regarding testing brain stimulation parameters (i.e., rTMS vs. iTBS) and individualizing coil placement for optimal targeting. We anticipate that active 10 Hz rTMS or iTBS will demonstrate target engagement compared to sham, and potentially ameliorate SCog deficits in people with SSDs. Our primary goal is to identify which treatment best induces change in SCog brain circuitry and secondarily which treatment is best tolerated and induces changes in social cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 years;
2. Male or Female;
3. DSM-5 diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder; other specified psychotic disorder (documented by SCID-5);
4. Prescription of antipsychotic medication for at least 60 days and constant dose for 30 days prior to study entry (either first or second generation antipsychotics permitted);
5. Able to participate in the informed consent process and provide voluntary informed consent.

Exclusion Criteria:

1. DSM-5 substance use disorder (other than caffeine, mild cannabis use, or tobacco) within the past six months; or a positive baseline urine drug screen (except cannabis for mild use). Only participants meeting a moderate to severe cannabis use disorder will be excluded
2. Type 1 diabetes mellitus (i.e., insulin-dependent diabetes mellitus with onset < 35 years of age and/or diabetes mellitus that has been complicated by a prior documented episode of ketoacidosis)
3. Acute or unstable medical illness (e.g. delirium, cancer, uncontrolled diabetes, decompensated cardiac, hepatic, renal or pulmonary disease, stroke, or myocardial infarction), whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol
4. Neurological disease associated with extrapyramidal signs and symptoms (e.g. Parkinson's disease); epilepsy (i.e. seizures not due to medication/drugs or due to fever) or physical signs of stroke; any diagnosis of a Central Nervous System (CNS) disorder
5. Requires a benzodiazepine with a regular dose equivalent to lorazepam 2 mg/day or higher or any anticonvulsant due to the potential of these medications to limit the efficacy of rTMS
6. Suspected DSM-5 intellectual disability based upon clinical interview and psychosocial history or estimated IQ of <71
7. Prior Psychosurgery
8. Presence of MRI contraindications (e.g. pacemakers)
9. Pregnancy (self-report)
10. rTMS treatment in the last 5 years
11. Non-English speakers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Change in mentalizing brain network functional connectivity | 2 weeks
  Measured using the empathic accuracy fMRI task

SECONDARY OUTCOMES:
Treatment Tolerability | 2 weeks
  Measured using the Visual Analogue Scale for Pain (VAS)
Treatment Tolerability | 2 weeks
  Measured using proportion of participants that report headache
Treatment Tolerability | 2 weeks
  Measured using proportion of participants that report dizziness
Treatment Tolerability | 2 weeks
  Measured using proportion of treatment related SAE's

CONTACTS AND LOCATIONS:
Overall Officials: Aristotle Voineskos, MD, Principal Investigator — Centre for Addiction and Mental Health; Anil Malhotra, MD, Principal Investigator — The Feinstein Institute for Medical Research, Zucker Hillside Hospital; Robert Buchanan, MD, Principal Investigator — Maryland Psychiatric Research Centre, University of Maryland
Locations (3):
- United States (2):
  - Maryland Psychiatric Research Centre, Catonsville, Maryland
  - The Feinstein Institute for Medical Research, Manhasset, New York
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes